CLINICAL TRIAL: NCT03201471
Title: Chidamide With R-CHOP Regimen for de Novo, High Risk Diffuse Large B Cell Lymphoma (DLBCL): A Prospective, Signal Arm, Open Label Clinical Trial
Brief Title: Chidamide With R-CHOP Regimen for DLBCL Patients
Acronym: DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Wenbin Qian, Chief of lymphoma center, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lymphoma center Q001
Record Dates: First submitted 2017-06-23; First posted 2017-06-28 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; HBI-8000

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): In this group, the patients will receive 2 courses of Chidamide+ R-CHOP regimen, the way of administration and dosage of the medicine used in the trial is as follows: Rituximab 375mg//m2, ivgtt,d1; CTX 750mg/m2, ivgtt,d2; EPI 70mg/m2, ivgtt,d2; VCR 1.4 mg/m2, ivgtt, d2; Pred 60 mg/m2, PO, d2-6; Chidamide 20mg/d,d1、4、8、11、14、18; one cycle every 21 days； abbreviation： CTX： cyclophosphamide；EPI：etoposide；VCR： vincristine；Pred：prednisone； R-CHOP：the chemo-therapy regimen composed of Rituximab, cyclophosphoamide; etoposide, vincristine and prednisone.
  Interventions: Drug: Chidamide + R-CHOP regimen

INTERVENTIONS:
Drug: Chidamide + R-CHOP regimen — Patients will receive 2 courses of Chidamide+ R-CHOP regimen, the way of administration and dosage of the medicine used in the trial is as follows: Rituximab 375mg//m2, ivgtt,d1;CTX 750mg/m2, ivgtt,d2;EPI 70mg/m2, ivgtt,d2;VCR 1.4 mg/m2, ivgtt, d2; Pred 60 mg/m2,PO, d2-6; Chidamide 20mg/d,d1、4、8、11、14、18;one cycle every 21 days;
  Other Names: HBI-8000

SUMMARY:
It's a prospective, single arm, open label phase II clinical trial, in which the safety and efficacy of Chidamide plus R-CHOP regimen is accessed in de novo DLBCL patients, who have received 2 courses of R-CHOP but only achieved PR or whose MRD tests for ctDNA revealed positive results.

abbreviation: R-CHOP: the chemo-therapy regimen composed of Rituximab, cyclophosphoamide, etoposide, vincristine and prednisone.

PR: partial remission; MRD:minimal residual disease;

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as diffuse large B-cell Lymphoma with positive CD20 results;
2. Age between 18 to 75 years old;
3. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) 0-2;
4. No history of malignant tumors, having no tumor other than DLBCL at the time of enrollment;
5. Life expectancy no less than 6 months
6. The patient or his/her attorney would be able to provide written consent for necessary examinations or procedures;
7. IPI mark>1.

Exclusion Criteria:

1. History of autologous stem cell transplantation;
2. History of other malignant tumors, except skin basal cell carcinoma and in situ cervical cancer;
3. With uncontrolled cardiovascular/ cerebrovascular disease, coagulation disorders, connective tissue disease, severe infectious diseases;
4. Lymphoma originated in the central nervous system;
5. Left ventricular ejection fraction ≦50％
6. Abnormal lab results in enrollment:

   1. Neutrophil count: <1.5*109/L；
   2. Platelet count <75*109/L；
   3. AST or ALT >2 times the upper limit of normal level，AKP and total bilirubin >1.5 times the upper limit of normal level;
   4. serum creatinine >1.5 times the upper limit of normal level;
7. Other uncontrolled medical conditions which the investigators think might influence the results of the trial;
8. Patients with mental illnesses or other diseases that might not comply with the trial plan;
9. Women during pregnancy or lactation;
10. HIV positive patients;
11. HbsAg (+) patients with HBV DNA(+), can be enrolled only when his/her HBV DNA turns negative; patients with HBsAg(-) HBcAb(+) can be enrolled only when his/her HBV DNA turns negative;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-02-05 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | every 3 months until 30 months after the last patient's enrollment
  complete remission rate after treated by Chidamide+ R-CHOP regimen

SECONDARY OUTCOMES:
progression free survival | from the day of treatment to the date of first documented progression，up to 30 months after the last patient's enrollment
  from date of inclusion to date of progression, relapse, or death from any cause
overall survival | 30 months after the last patient's enrollment
  from the date of inclusion to date of death, irrespective of cause
adverse events | from the date of first cycle of treatment to 30 months after last patient's enrollment
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
All the data would be available on the corresponding website of the leading research center.